CLINICAL TRIAL: NCT00003560
Title: A Phase II Study of Docetaxel and Carboplatin for Suboptimally Debulked Stage III or Stage IV Ovarian and Fallopian Tube Carcinoma
Brief Title: Docetaxel Plus Carboplatin in Treating Patients With Stage III or Stage IV Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Herbert Irving Comprehensive Cancer Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066624; CPMC-IRB-8437; NCI-V98-1467
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2003-09

CONDITIONS: Endometrial Cancer; Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; stage III endometrial carcinoma; stage IV endometrial carcinoma; endometrial papillary serous carcinoma; fallopian tube cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Endometrial Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Carboplatin; Docetaxel

INTERVENTIONS:
Drug: carboplatin
Drug: docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining docetaxel and carboplatin in treating patients who have stage III or stage IV ovarian cancer, fallopian tube cancer, or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the response rate, duration of response, and progression-free and overall survival of previously untreated patients with suboptimally debulked stage III or stage IV ovarian carcinoma, fallopian tube carcinoma, papillary serous cancer of the uterus, or primary peritoneal carcinoma treated with docetaxel and carboplatin.
* Evaluate the feasibility and toxicity of this regimen in these patients.
* Evaluate the effect of this regimen on quality of life of these patients.

OUTLINE: This is an open-label study.

Patients receive docetaxel IV over 1 hour and carboplatin IV over 30 minutes on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed prior to therapy and then after every 3 courses of chemotherapy.

PROJECTED ACCRUAL: Approximately 14-40 patients will be accrued for this study within 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed previously untreated ovarian cancer, fallopian tube carcinoma, papillary serous cancer of the uterus, or primary peritoneal carcinoma

  * Suboptimally debulked stage III or suboptimally or optimally debulked stage IV
* Measurable or evaluable disease

  * CNS lesions, lytic bone lesions, and radiated lesions (unless there is documented progression after radiotherapy) are not considered measurable
  * CA 125 levels above 49 units/mL in the absence of cirrhosis or nonmalignant gross ascites are considered evaluable
* Ineligible for other high-priority national or institutional study

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* ECOG 0-1

Life expectancy:

* More than 2 months

Hematopoietic:

* WBC greater than 3,000/mm3
* Platelet count greater than 100,000/mm3

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* SGOT and/or SGPT less than 2.5 times ULN OR
* SGOT and/or SGPT no greater than 2.5 times ULN if alkaline phosphatase no greater than ULN OR
* Alkaline phosphatase no greater than 4 times ULN if SGOT and/or SGPT no greater than ULN
* No SGOT and/or SGPT greater than 1.5 times ULN with alkaline phosphatase greater than 2.5 times ULN
* Alkaline phosphatase less than 350 U/L

Renal:

* BUN less than 1.5 times normal
* Creatinine less than 1.5 times ULN

Other:

* No other malignancy within the past 5 years except curatively treated carcinoma in situ of the cervix or skin cancer
* No other serious medical or psychiatric illness
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormone therapy

Radiotherapy:

* See Disease Characteristics
* No prior radiotherapy

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 1998-05

CONTACTS AND LOCATIONS:
Overall Officials: Amy D. Tiersten, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (1):
- Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York, United States